CLINICAL TRIAL: NCT06853236
Title: A Cardiorespiratory Fitness Test for Acute Illness: Validity, Reliability, and Clinical Utility of Functional Incremental Stepping-in-Place Test
Brief Title: Functional Incremental Stepping in Place Test (F-IST) Validation
Acronym: F-IST
Status: Recruiting | Type: Observational
Sponsor: Kirby Mayer (Other)
Collaborators: Duke University (Other); Florida Atlantic University (Other)
Responsible Party: Sponsor-Investigator, Kirby Mayer, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 86390; 1000400362 (Other Grant/Funding Number: Foundation for Physical Therapy)
Record Dates: First submitted 2025-02-14; First posted 2025-02-28 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Intensive Care Medicine; Acute Care Medical
Keywords: Cardio respiratory fitness; incremental step test; validity; reliability; physical function; graded exercise testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy: Community-dwelling older adults (≥60 years) with no recent hospitalization
- ICU Survivor: Patients who survived ICU admission for ARF or sepsis in the last year
- Chronic Pulmonary Disease: Community-dwelling adults with diagnosis of COPD, ILD, or PF

SUMMARY:
The purpose of this multi-site prospective study is to assess validity of a new step test called Functional-Incremental Stepping-in-place- Test (F-IST) compared to gold-standard cardiopulmonary exercise testing (CPET) and to physical function and health perception, respectively. The investigators will also assess test-retest reliability of the F-IST. The investigators hypothesize that the F-IST will have high validity and test-retest reliability to be used in field testing environments such as the ICU.

DETAILED DESCRIPTION:
Acutely hospitalized patients are at risk for hospital-acquired functional decline (HAD). This decline increases the likelihood of developing physical disability after discharge, particularly in those with older age, multimorbidity, pre-existing functional impairment and life support exposures (i.e. mechanical ventilation). Identifying patients at increased risk provides important prognostic data to inform planning strategies for both in-hospital and post-acute intervention.

Common physiological consequences associated with HAD are diminished skeletal muscle function and cardiorespiratory fitness (CRF). Historically, the six-minute walk test (6MWT) has been utilized as a chief outcome measure in the acute hospitalization and post-discharge phases to examine functional exercise capacity, estimate maximal capacity, and prescribe exercise intervention. The 6MWT is a submaximal field test that allows patients to self-select their walking pace and may be influenced by several factors including motivation. The internally-selected pace coupled with the lack of incremental increases in intensity can underrepresent CRF. In addition, the test requires a 30-meter straight course, which can be challenging to find in the hospital environment. Thus, to address the limitations of submaximal field tests, our team developed the Functional-Incremental Stepping-in-place Test (F-IST).

Designed to objectively examine CRF across the variety of patients encountered in clinical practice, the F-IST is an incremental, externally-paced, symptom-limited stepping-in-place test. While maintaining the graded components of gold standard cardiopulmonary exercise testing (CPET), it has high clinical utility since it requires minimal equipment (UE support allowed), minimal space (performed at bedside), and short administration time (< 10 min). Also, the incremental increase in intensity is individualized to perceived exertion and heart rate responses during test stages, which ultimately enables precise exercise prescription. Preliminary data on F-IST from the ongoing randomized controlled trial (NCT05218083) demonstrate potential for strong construct validity when compared to 6MWT (n = 9, spearman rho = 0.65, p = 0.05). However, before implementation in clinical practice, a new test requires the study of its measurement properties to assure that its selection is evidence-based.

Findings from this study will demonstrate that F-IST is a robust valid and reliable assessment of CRF that can be implemented on the frontline of acute care physical therapy. The F-IST addresses important limitations of field tests with an enhanced rigor by maintaining principles of gold-standard CPET. The F-IST will enable clinicians and researchers to provide precision exercise prescription to optimize patient function.

ELIGIBILITY:
Inclusion Criteria:

-Currently able to walk with or without a walking aid, such as a cane or walker or rollator

Exclusion Criteria:

Pregnancy

specifically related to cardiopulmonary testing

* A recent significant change in resting ECG
* Unstable angina
* Uncontrolled cardiac dysrhythmias causing symptoms or hemodynamic compromise
* Symptomatic severe aortic stenosis
* Uncontrolled symptomatic heart failure
* Acute pulmonary embolus or pulmonary infarction
* Acute myocarditis or pericarditis
* Suspected or known dissecting aneurysm
* Acute systemic infection accompanied by fever, body aches, or swollen lymph glands
* Left Main Coronary Stenosis
* Moderate stenotic valvular heart disease
* Electrolyte abnormalities
* Severe arterial hypertension (>200 systolic, >110 diastolic) at rest
* Tachydysrhythmia or bradydysrhythmia
* Hypertrophic cardiomyopathy and other forms of outflow tract obstruction
* Neuromuscular, musculoskeletal, or rheumatic disorders that are exacerbated by exercise
* High degree AV block
* Ventricular aneurysm
* Uncontrolled metabolic disease (diabetes, thyrotoxicosis, or myxedema)
* Chronic infectious disease (hepatitis, AIDS, mono)
* Mental or physical impairment leading to inability to exercise adequately

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This project may include adults aged 18 and older without regard to sex, race, or ethnicity. Exclusions will include pregnancy and vulnerable groups such as children, prisoners, adults with impaired consent capacity or are non-English speaking. All participation must be on a voluntary basis.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Modified Bruce Treadmill VO2 Peak | Upon enrollment at baseline (day 0-7)
  Peak oxygen consumption during the modified Bruce cardiorespiratory test using a PARVO metabolic cart
F-IST VO2 Peak | Upon enrollment at baseline (day 0-7)
  Peak oxygen consumption during the F-IST cardiorespiratory test using a PARVO metabolic cart
F-IST VO2 Peak Reliability | Approximately 1-2 weeks following baseline (day 14-21)
  Peak oxygen consumption during the F-IST cardiorespiratory test using a PARVO metabolic cart

SECONDARY OUTCOMES:
6MWT distance | Approximately 1-2 weeks following baseline (day 14-21)
  Six minute walking test distance in meters
4m habitual gait speed | Approximately 1-2 weeks following baseline (day 14-21)
  Habitual gait speed across a 4 meter distance
Sit to Stand Test (5x) | Approximately 1-2 weeks following baseline (day 14-21)
  Time in seconds it takes to rise and sit from a chair 5 times
Sit to Stand Test (30 seconds) | Approximately 1-2 weeks following baseline (day 14-21)
  The number of full repetitions completed to rise and sit from a chair over 30 seconds
EQ5D-5L Questionnaire | Approximately 1-2 weeks following baseline (day 14-21)
  Health related quality of life scale patient reported outcome
Visual Analog Scale Questionnaire | Approximately 1-2 weeks following baseline (day 14-21)
  Health related quality of life scale patient reported outcome
FACIT-fatigue Questionnaire | Approximately 1-2 weeks following baseline (day 14-21)
  Patient reported outcome indicating fatigue
SF-36 Questionnaire | Approximately 1-2 weeks following baseline (day 14-21)
  Patient reported outcome indicating eight different domains of health
St. George's Respiratory Questionnaire | Approximately 1-2 weeks following baseline (day 14-21)
  Patient reported outcome measuring impact of overall health, daily life, and respiratory systems

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Florida Atlantic University, Boca Raton, Florida
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
The dissemination plan emphasizes transparency of the study, and as a study team, the investigators are committed to sharing de-identified data for external researchers.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: IPD will be available at the time of manuscript acceptance and publishing. A published manuscript is planned for late 2026.
Access Criteria: Any external researcher will be able to access de-identified, non, PHI, individual participant data as part of the journal's supplementary information.